CLINICAL TRIAL: NCT00341328
Title: Efficacy and Safety of Immunomodulator (Mycobacterium w.) as an Adjunct Therapy in Category I Pulmonary Tuberculosis and Along With Assessment of Immunological Parameters
Brief Title: Efficacy and Safety of Immunomodulator as an Adjunct Therapy in New Pulmonary Tuberculosis(Category I) Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, SK Sharma, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-01C-1/2003-10; BT/PR7894/Med/14/1175/2006 (Other: Department of Biotechnology, MST, India)
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Tuberculosis
Keywords: India; Pulmonary Tuberculosis; Category-I Pulmonary Tuberculosis; Immunomodulator; Mycobacterium w
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Immuvac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In one arm the patient will receive intradermal Mycobacterium W Vaccine along with Category I ATT drugs according to RNTCP guidelines
  Interventions: Biological: Intradermal injection of Mycobacterium w
- 2 (Placebo Comparator): In this Arm patient will receive Placebo along with Category I ATT drugs according to RNTCP guidelines
  Interventions: Biological: Intradermal injection of Mycobacterium w

INTERVENTIONS:
Biological: Intradermal injection of Mycobacterium w — Mw Vaccine is given as intradermal administration. Total 6 doses are given 0.2 ml at baseline and then 0.1 ml after interval of 2 weeks upto 8 weeks
  Other Names: Immuvac

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Mycobacterium w in new lung tuberculosis patients. Mycobacterium w is a strain of bacterium which is being used as vaccine and adjunct drug against leprosy. This agent has also been found to be useful in the treatment of lung tuberculosis in limited number of patients.

We are conducting this study in category-I patients( As per World Health Organization,Geneva classification of tuberculosis) having lung tuberculosis to see the efficacy and also to see any change in the immunological parameters.

DETAILED DESCRIPTION:
Mycobacterium w is a recently introduced immunomodulator ,which has been found to be useful in rapid killing of Mycobacterium leprae. It improves clearance of Mycobacterium leprae from body and is thereby useful in reducing duration of therapy significantly for multibacillary leprosy. Mycobacterium w shares antigens with Mycobacterium leprae as well as Mycobacterium tuberculosis. Mycobacterium w is also found to be useful in prevention of tuberculosis in experimental animals. Previous studies for efficacy of Mycobacterium w as immunomodulator in pulmonary tuberculosis patients have shown faster sputum conversion rates in patients given Mycobacterium w as an adjuvant therapy along with standard anti-tuberculosis treatment. It has faster and remarkable sputum converting capacity. Similar studies conducted in pulmonary TB category -II [Re-treatment as per Revised National Tuberculosis Control Programme (RNTCP), Govt. of India] patients have shown improved cure rates.

Mycobacterium w is commercially available under the brand name of "Immuvac" injection in 0.5 ml multi-dose vials approved for use as immunomodulator against Mycobacterium leprae in patients with leprosy. Each vial has 500 million heat-killed bacilli in a buffered solution. It is manufactured by Cadila Pharmaceuticals Ltd.; Ahmedabad, Gujarat-382 210, India. In this clinical trial one dose consists of 0.1 ml given as intradermal injection, which contains 100 million bacilli. A total of 6 doses are given during the Intensive Phase(as per RNTCP,Ministry of Health and Family Welfare,Govt.of India) of treatment. Two injections on both upper arms on day-0 and subsequently one injection on days 14,28,42 and 56. No injections are given during the Continuation Phase(as per RNTCP,Ministry of Health and Family Welfare,Govt.of India)of treatment.

As of now it is not commercially available for therapeutic use in TB patients as immunomodulator.Therefore we are investigating Mycobacterium w for its efficacy in TB patients in a "double-blind placebo-controlled randomized clinical control trial" fashion. We are conducting this trial in Category-I pulmonary TB Patients(as per RNTCP,Ministry of Health and Family Welfare,Govt.of India),and are assessing the outcome in the form of clinical improvement,sputum conversion and immunological parameters. This is a multi-centric trial sponsored by the Department of Biotechnology, Ministry of Science and Technology, Govt. of India and Cadila Pharmaceuticals Ltd., India.

ELIGIBILITY:
Inclusion Criteria

1. Patients of either sex aged between 18 to 60 yrs.
2. Newly diagnosed sputum positive pulmonary TB cases with at least 2 sputum samples that are positive on sputum microscopy (Negative, Scanty, Scanty may be enrolled.
3. Patients who are willing to give an informed consent.

Exclusion Criteria

1. Known hypersensitivity to Category I anti-TB drugs on history at the time of Screening.
2. Known history of DR-TB (includes MDR-TB and XDR-TB) at the time of screening. Patients with Mtb isolate resistant to one or more drugs are to be excluded.
3. Presence of secondary immunodeficiency states: HIV, organ transplantation, diabetes mellitus, malignancy, treatment with corticosteroids (illicited on detailed history and lab investigations).
4. Hepatitis B and C positivity.
5. Patients with known extrapulmonary TB and/or patients requiring surgical intervention.
6. Currently receiving cytotoxic therapy, or have received it within the last 3 months- Ask on History.
7. Pregnancy and lactation on history.
8. Patients with a known seizure disorder on history.
9. Patients with known symptomatic cardiac disease, such as arrhythmias or coronary artery disease on history.
10. Patients with abnormal renal function (Serum creatinine more than 1.5 or proteinuria more than 2+ )
11. Patients with abnormal hepatic functions (bilirubin = 1.5 mg/dl; AST, ALT, SAP more than 1.5 x ULN; PT = 1.3x control)
12. Patients with hematological abnormalities (WBC lesser than or equal to 3000/mm3; platelets less than or equal to 100,000/mm3).
13. Seriously ill and moribund patients with complications:

    1. low lung reserve, marked tachypnoea, chronic cor pulmonale, congestive cardiac failure, BMI<15,
    2. severe hypoalbuminemia (< 2.5 g/dl).
14. Patients unlikely to survive for less than 6 months.
15. Patients unable to comply with the treatment regimen.
16. Patients with history of alcohol or drug abuse- to be asked for on history and assessed using the CAGE Questions. The patient should be asked four questions in the following manner. A positive response to any of the following questions will be considered an exclusion criterion.

    i. Have you ever felt a need to CUT DOWN your drinking?

    ii. Have you ever felt ANGRY when confronted about the amount of alcohol you drink?

    iii. Have you ever felt GUILTY when confronted about the amount of alcohol you drink?

    iv. Have you ever felt the need to have a drink first thing in the morning? (EYE OPENER).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2007-03; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The time of sputum conversion as well as the early sputum conversion between the two groups will be evaluated. | from the baseline(visit 2)
The cure rate will be evaluated as the primary parameter of efficacy. | 6-7 month
The relapse in patients of category-I pulmonary TB will be compared in both the groups. | at an interval of 6,12,18 and 24 months after the completion of the therapy
Recording of any clinical adverse reactions for assessment of safety. | at anytime during the study

SECONDARY OUTCOMES:
An additional secondary efficacy endpoint is the patient's and physicians's global assessment of the clinical cure. | 6-7 month

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, Ph.D., Study Chair — Professor and Head,Department of Medicine, AIIMS, New Delhi-110029; Bindu Dey, Ph.D., Study Director — Department of Biotechnology, MST, GOI
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Central JALMA Institute of Leprosy and Other Mycobacterial Diseases, Agra

REFERENCES:
- [Background] Patel N, Trapathi SB. Improved cure rates in pulmonary tuberculosis category II (retreatment) with mycobacterium w. J Indian Med Assoc. 2003 Nov;101(11):680, 682. PMID 15198421
- [Background] Patel N, Deshpande MM, Shah M. Effect of an immunomodulator containing Mycobacterium w on sputum conversion in pulmonary tuberculosis. J Indian Med Assoc. 2002 Mar;100(3):191-3. PMID 12408283
- [Background] Katoch K, Katoch VM, Natrajan M, Bhatia AS, Sreevatsa, Gupta UD, Sharma VD, Shivannavar CT, Patil MA, Bharadwaj VP. Treatment of bacilliferous BL/LL cases with combined chemotherapy and immunotherapy. Int J Lepr Other Mycobact Dis. 1995 Jun;63(2):202-12. PMID 7602215
- [Background] Sharma P, Mukherjee R, Talwar GP, Sarathchandra KG, Walia R, Parida SK, Pandey RM, Rani R, Kar H, Mukherjee A, Katoch K, Benara SK, Singh T, Singh P. Immunoprophylactic effects of the anti-leprosy Mw vaccine in household contacts of leprosy patients: clinical field trials with a follow up of 8-10 years. Lepr Rev. 2005 Jun;76(2):127-43. PMID 16038246
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Disabilities in multibacillary leprosy following multidrug therapy with and without immunotherapy with Mycobacterium w antileprosy vaccine. Int J Lepr Other Mycobact Dis. 1999 Sep;67(3):250-8. PMID 10575404
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Reactional states and neuritis in multibacillary leprosy patients following MDT with/without immunotherapy with Mycobacterium w antileprosy vaccine. Lepr Rev. 2000 Jun;71(2):193-205. doi: 10.5935/0305-7518.20000021. PMID 10920614
- [Background] Sharma P, Misra RS, Kar HK, Mukherjee A, Poricha D, Kaur H, Mukherjee R, Rani R. Mycobacterium w vaccine, a useful adjuvant to multidrug therapy in multibacillary leprosy: a report on hospital based immunotherapeutic clinical trials with a follow-up of 1-7 years after treatment. Lepr Rev. 2000 Jun;71(2):179-92. doi: 10.5935/0305-7518.20000020. PMID 10920613
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Induction of lepromin positivity following immuno-chemotherapy with Mycobacterium w vaccine and multidrug therapy and its impact on bacteriological clearance in multibacillary leprosy: report on a hospital-based clinical trial with the candidate antileprosy vaccine. Int J Lepr Other Mycobact Dis. 1999 Sep;67(3):259-69. PMID 10575405
- [Background] Sharma SK, Mitra DK, Balamurugan A, Pandey RM, Mehra NK. Cytokine polarization in miliary and pleural tuberculosis. J Clin Immunol. 2002 Nov;22(6):345-52. doi: 10.1023/a:1020604331886. PMID 12462334
- [Background] Khatri GR, Frieden TR. Controlling tuberculosis in India. N Engl J Med. 2002 Oct 31;347(18):1420-5. doi: 10.1056/NEJMsa020098. PMID 12409545